CLINICAL TRIAL: NCT02308384
Title: The Use of Immunochemical Faecal Occult Blood Test (iFOBT) in General Practice. A Randomised Trial of the Implementation of iFOBT.
Brief Title: A Trial of the Implementation of iFOBT in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Randomiseret iFOBT studie
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2015-11

CONDITIONS: Colorectal Cancer
Keywords: iFOBT; FIT; general practice; early diagnosis
MeSH Terms: conditions — Colorectal Neoplasms; Disease | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Before intervention (No Intervention): GPs in this group have not yet received intervention.
- After intervention (Experimental): GPs in this group have received the intervention.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — CME, Start-package and status mail
  Arms: After intervention

SUMMARY:
Background

Colorectal cancer (CRC) is common, and a leading cause of cancer death. The evaluation of patients suspected to have CRC is difficult due to poorly predictive alarm symptoms and many patients present with uncharacteristic or vague symptoms. The faecal marker of human globin, iFOBT, could play an important role in aiding the general practitioner in detecting CRC.

Hypothesis

It will be possible to implement iFOBT in general practice as a test performed on patients who do not fulfill the criteria for fast-track referral for colorectal cancer, but whose symptoms could indicate an undiagnosed colorectal cancer.

Aim

To implement iFOBT in general practice and evaluate the uptake and clinical use of the test. Furthermore, we want to investigate the performance of iFOBT when used on patients presenting with uncharacteristic symptoms of CRC, and the clinical implications.

Materials and methods

The study uses a cluster randomised stepped wedge design. Clusters are constituted by the 18 municipalities in the central Denmark Region, and these are randomised when to receive a continuous medical education (CME). The date of inclusion is defined as the first working day in the month the CME is planned to be conducted. The CME is part of an intervention aimed to facilitate the implementation of iFOBT in general practice. Besides a CME, the intervention consist of a start package (iFOBT kits, a guideline and online educational material) that is sent to GPs when they are included in the study, and a status mail that GPs receive approx. one month after inclusion. The inclusion period is during the first 7 month of the study period, the study lasts for one year.

Perspectives

This study will provide important knowledge on how to improve CRC diagnostics in general practice.

DETAILED DESCRIPTION:
Background

Colorectal cancer (CRC) is the second most common type of cancer in Denmark and is a leading cause of cancer death. Since 2000, the incidence has been increasing by 1-1.5% each year. The estimated 5-year survival rate is currently 80% for stage I cancer, 50% for stages II and III, and <5 % for stage IV cancer. These figures emphasize the importance of detecting the disease in early stages and underline the current challenge of diagnosing CRC in general practice.

In 2008, a national fast-track system for cancer patients was established to ensure fast diagnosis and initiation of treatment. The fast-track system implies that patients presenting 'alarm' symptoms of e.g. CRC will be referred immediately for diagnostic workup; no more than 14 days must pass from referral to initiation of treatment. Several studies have shown that the positive predictive values (PPV) of the symptoms regarding CRC are fairly low (4-8%). In addition, approximately 50% of new CRC incidents will present with other vague and uncharacteristic symptoms than alarm symptoms.

In addition, a screening programme for CRC has been implemented. It is suggested that this will increase survival rate of CRC, however, it is estimated that approximately 75% of yearly CRC still have to be diagnosed through general practice.

A huge load is, consequently, still placed on general practice in the quest for earlier diagnosis of CRC, and better methods to aid the general practitioner in the diagnostic process are needed.

One tool could be the use of iFOBT in general practice for patients who present with symptoms that could origin from an underlying CRC, but without being alarm symptoms.

Aim

To implement iFOBT in general practice and evaluate the uptake and clinical use of the test. Furthermore, we want to investigate the performance of iFOBT when used on patients presenting with uncharacteristic symptoms of CRC, and the clinical implications.

Materials and methods

We will develop a guideline for the use of iFOBT in general practice. The guideline is aimed at men and women aged 30 years and above who present symptoms that could origin from a CRC, but are not classified as alarm symptoms. The guideline will contain a list of symptoms for which it is recommended to perform iFOBT and suggested actions for positive and negative test result. A value of <49µg/L will be considered 'negative' and >50µg/L as 'positive'.

The study uses a cluster randomised stepped wedge design, and is executed in the Central Denmark Region. Municipalities of the region are randomised when to receive a CME, and are included sequentially in the study during the first seven month of the study period. The CME are arranged on scheduled GP-meetings in each municipality and will consist of a 45 minutes lecture on CRC diagnosis and use of iFOBT. Besides a CME, the intervention consist of a start package (10 iFOBT kits, a guideline and online educational material) that is sent to GPs when they are included in the study, and a status mail that GPs receive approx. one month after inclusion. The study period is one year. Data analysis will focus on the uptake and clinical use of iFOBT in general practice, the performance of iFOBT when used on patients presenting with uncharacteristic symptoms of CRC and the clinical implications.

Perspectives

This study will investigate iFOBT and explore its role in general practice. To our knowledge, this study will be one of the first and most thorough investigations of this test in a primary care setting. The results will bring important knowledge of how to improve the diagnostics of colorectal cancer in the future and hopefully reduce time to diagnosis. Especially for patients who do not meet the traditional Danish criteria for fast-track referral, this study will be a corner stone in the identification of more efficient ways to locate patients at risk of developing CRC. At both national and international level, this project will contribute with important knowledge that may provide better planning of CRC diagnostics in the future.

ELIGIBILITY:
Inclusion Criteria:

* GPs in the Central Denmark Region
* Patients >30 years eligible for iFOBT according to guideline

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The rate of positive iFOBTs | 1 year
The number of CRCs diagnosed after a positive iFOBT | 1 year
The stage distribution of CRCs for patients with a positive iFOBT | 1 year
  UICC stages I-IV
The positive predictive value for detecting colorectal cancer | 1 year
  The risk of having CRC when the iFOBT is positive
The positive predictive value for detecting colorectal cancer in relation to cut-off value of iFOBT | 1 year
  The risk of having CRC at different iFOBT values.
The positive predictive value for detecting colorectal cancer in relation to indications of using iFOBT | 1 year
  The risk of having CRC when iFOBT is positive and specific symptoms. When requesting FIT, the GP register the patients' symptoms.

SECONDARY OUTCOMES:
The rate of general practices starting to use the iFOBT, stratified for participation in the CME. | 1 year
  The relation between number of general practices started using iFOBT and time.
The monthly rate of requested iFOBTs, stratified for participation in the CME. | 1 year
  The relation between number of requested iFOBTs and time.
The monthly rate of positive iFOBTs, stratified for participation in the CME. | 1 year
  The relation between number of positive iFOBTs and time.
Indications used for requesting iFOBT, stratified for participation in the CME. | 1 year
The rate of referrals in the cancer patient pathway for colorectal cancer | 1 year
The rate of performed colonoscopies | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vedsted, Professor, Study Director — Research Unit of General Practice, Odense
Locations (1):
- Research Unit for General Practice, Aarhus C, Denmark

REFERENCES:
- [Derived] Juul JS, Bro F, Hornung N, Andersen BS, Laurberg S, Olesen F, Vedsted P. Implementation of immunochemical faecal occult blood test in general practice: a study protocol using a cluster-randomised stepped-wedge design. BMC Cancer. 2016 Jul 11;16:445. doi: 10.1186/s12885-016-2477-9. PMID 27400657